CLINICAL TRIAL: NCT05120232
Title: Flourishing and Virtue in Cognitive-Behavioral Therapy for Anxiety and Depressive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: University of Kentucky (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61245; 5724E (Other: BU CRC IRB)
Record Dates: First submitted 2020-09-08; First posted 2021-11-15 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Anxiety Disorders; Depressive Disorder
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified Protocol (UP) (Active Comparator): The Unified Protocol (UP) is a transdiagnostic, cognitive-behavioral therapy that has been shown to be effective for treating emotional disorders. The UP targets negative emotions and helps people respond to their emotions in ways that are more helpful for them and in line with their goals. This will be delivered entirely on an online platform.
  Interventions: Behavioral: Unified Protocol
- Modified Unified Protocol (UP+) (Experimental): A modified version of the UP (called the UP+) delivered entirely on an online platform that will include exercises specifically designed to enhance positive emotions.
  Interventions: Behavioral: Modified Unified Protocol (UP+)

INTERVENTIONS:
Behavioral: Unified Protocol — A transdiagnostic, cognitive behavioral therapy.
  Arms: Unified Protocol (UP)
Behavioral: Modified Unified Protocol (UP+) — A transdiagnostic, cognitive behavioral therapy.
  Arms: Modified Unified Protocol (UP+)

SUMMARY:
This two phase study is testing an online version of a transdiagnostic, cognitive behavioral therapy, against a modified version of that therapy emphasizing positive affect. The first phase of the trial will focus on content development for the modified therapy and the second phase will be a randomized control trial comparing the two.

DETAILED DESCRIPTION:
Research shows that positive emotions can buffer against the effects of stress as well as contribute to overall well-being and functioning. People with emotional disorders, such as anxiety and depression, often report lower levels of positive emotions. However, to date, most existing treatment approaches for emotional disorders focus on regulating negative emotions, without explicitly focusing on positive emotions.

The Unified Protocol (UP) is a transdiagnostic, cognitive-behavioral therapy that has been shown to be effective for treating emotional disorders. The UP targets negative emotions and helps people respond to their emotions in ways that are more helpful for them and in line with their goals. In its current form, the UP does not explicitly target positive emotions, but some research suggests that individuals treated with the UP and other cognitive-behavioral treatments experience some improvement in positive affect.

In the current study, the researchers will create a modified version of the UP (called the UP+) delivered entirely on an online platform that will include exercises specifically designed to enhance positive emotions. Then, the researchers will evaluate the UP+ in a small sample of participants to examine acceptability and feasibility and will then use this information to continue to refine the protocol. Finally, the researchers will conduct a randomized controlled trial to assess the efficacy of the UP+. Participants diagnosed with emotional disorders will be randomized to either receive the UP or the UP+ delivered on an online platform and will be assessed on a range of outcomes, including positive and negative affect, psychological symptoms, and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with a DSM-5 anxiety, obsessive-compulsive, or depressive disorder

Exclusion Criteria:

Acute risk factors (suicidal or homicidal ideation or clinical condition requiring immediate treatment);

The individual is in treatment elsewhere for related issues; and/or

The individual is considering changing their treatment and and/or psychotropic medication during the time period in which they would be enrolled in the study and/or

The individual is unable or unwilling to commit to the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety and Related Disorders Interview Schedule for Diagnostic and Statistical Manual-5 (ADIS-5) Score | Baseline, 12-weeks following baseline, 3 months following the treatment phase
  This semi-structured, diagnostic clinical interview focuses on Diagnostic and Statistical Manual-5 diagnoses of anxiety disorders and their accompanying mood states, somatoform disorders, and substance and alcohol use. The information derived from the interview using the ADIS allows clinicians to determine differential diagnoses and gain a clear understanding of the level and severity of each diagnosis. Principal and additional diagnoses are assigned a clinical severity rating (CSR) on a scale from 0 (no symptoms) to 8 (extremely severe symptoms), with a rating of 4 or above (definitely disturbing/disabling) passing the clinical threshold for DSM diagnostic criteria. Inquiries about suicidal ideation are part of this interview. This measure has demonstrated excellent to acceptable interrater reliability for the anxiety and mood disorders (Brown, Di Nardo, et al., 2001).

OTHER OUTCOMES:
Change in Positive and Negative Affect Schedule Expanded Form (PANAS-X) Score | Baseline, every week through 12-weeks following baseline, 3 months following the treatment phase
  The PANAS-X is a brief, reliable and valid measure of positive and negative affect. It consists of 20 feeling or emotion words (e.g., interested, upset, nervous). Respondents rate each emotion word on a scale ranging from 1 = very slightly or not at all to 5 = extremely, indicating the extent to which they experience that emotion or feeling in general. The PANAS-X has shown excellent convergent and discriminant correlations with lengthier measures of underlying mood factors and is a widely used measure of state negative affect (Watson et al., 1988).
Change in Savoring Beliefs Inventory (SBI) Score | Baseline, every week through 12-weeks following baseline, 3 months following the treatment phase
  The SBI is a measure of one's tendency to savor or dampen positive emotions (Bryant, F. B. 2003). It includes distinctions among future, present, and past focused forms of savouring. The SBI includes 24 items with 4 positively-worded and 4 negatively-worded items for each of the three temporal forms of savoring (rated on a 7-point scale from 1 = strongly agree to 7 = strongly disagree) . Overall, the SBI is a valid and reliable measure of individuals' beliefs about their capacity to savour positive experiences (Bryant 2003).
Change in Flourish Index (FI) Score | Baseline, every week through 12-weeks following baseline, 3 months following the treatment phase
  The FI is a measurement approach to human flourishing, based around five central domains: happiness and life satisfaction, mental and physical health, meaning and purpose, character and virtue, and close social relationships. The FI consists of 10 questions on a 10 point Likert scale (with 0 = strongly disagree to 10 = strongly agree) (VanderWeele, 2017). The FI has demonstrated good internal consistency and evidence of validity and reliability (Węziak-Białowolska et al, 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Todd Farchione, Ph.D., Principal Investigator — Center for Anxiety Related Disorders at Boston University
Locations (1):
- Center for Anxiety and Related Disorders - Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teplow D, Spencer-Laitt D, Long LJ, Hey AJ, Moreno JD, Farchione TJ. Strengths use and emotional disorder symptom reduction during a transdiagnostic cognitive behavioral therapy: A random-intercept cross-lagged panel model study. Psychotherapy (Chic). 2025 Jun;62(2):220-234. doi: 10.1037/pst0000553. Epub 2024 Nov 21. PMID 39570688